CLINICAL TRIAL: NCT01074372
Title: A Randomized, Double-Blind,Placebo-Controlled, Ascending Single-Dose Study of the Safety, Tolerability and Bioeffect of Subcutaneously Administered REGN727 in Healthy Volunteers
Brief Title: Ascending Dose Study of the Safety and Tolerability of REGN727 (SAR236553) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R727-CL-0904
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Dose 1 versus placebo
  Interventions: Drug: REGN727; Drug: Placebo
- Cohort 2 (Experimental): Dose 2 versus placebo
  Interventions: Drug: REGN727; Drug: Placebo
- Cohort 3 (Experimental): Dose 3 versus placebo
  Interventions: Drug: REGN727; Drug: Placebo
- Cohort 4 (Experimental): Dose 4 versus placebo
  Interventions: Drug: REGN727; Drug: Placebo

INTERVENTIONS:
Drug: REGN727 — 4 cohorts (dose 1, 2, 3, 4)
Drug: Placebo — 4 cohorts (dose 1, 2, 3, 4)

SUMMARY:
This study will test the safety and tolerability (how the body reacts to the drug) of REGN727 compared with placebo (an inactive substance that contains no medicine) in healthy subjects. The study drug and placebo will be administered by an injection under the skin at one clinic visit. There will be 14 clinic visits, which will include 4 overnight stays. Subjects will be monitored by the study staff for side effects and the body's response to the study drug. Vital signs (blood pressure, temperature, breathing and heart rate) will be checked, and blood and urine samples will be collected at some or all visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 65 years of age.
* Weight> 50 kg and <95 kg inclusive
* For women of childbearing potential, a negative serum pregnancy test at the screening visit and a negative urine pregnancy test on day 1.
* For men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner[s] become pregnant during the full duration of the study.
* Willing, committed, and able to return for all clinic visits and complete all study-related procedures.
* Able to read, understand and willing to sign the informed consent form.

Exclusion Criteria:

* Initiation of a new exercise routine or major change to a previous exercise routine within 4 weeks prior to screening visit.
* Pregnant or breast-feeding females.
* Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease, or any other illness or condition that would adversely affect the subject's participation in this study.
* Hospitalization for any reason within 60 days of screening.
* Known history of Human Immunodeficiency Virus (HIV) antibody; and/or positive Hepatitis B surface antigen, and/or positive Hepatitis C antibody at the screening visit.
* Previous exposure to any therapeutic or investigational biological agent.
* History of alcohol or substance abuse within previous 5 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events in subjects treated with REGN727 or placebo, reported from the administration of study drug on day 1 to the completion of the study on day 106 | 106 days

CONTACTS AND LOCATIONS:
Overall Officials: Gary Swergold, MD, PhD, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Overland Park, Kansas, United States

REFERENCES:
- [Derived] Stein EA, Mellis S, Yancopoulos GD, Stahl N, Logan D, Smith WB, Lisbon E, Gutierrez M, Webb C, Wu R, Du Y, Kranz T, Gasparino E, Swergold GD. Effect of a monoclonal antibody to PCSK9 on LDL cholesterol. N Engl J Med. 2012 Mar 22;366(12):1108-18. doi: 10.1056/NEJMoa1105803. PMID 22435370